CLINICAL TRIAL: NCT06285994
Title: Complications of High Frequency Jet Ventilation During Bronchoscopy - a Retrospective Cohort Study
Brief Title: Complications of High Frequency Jet Ventilation
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SRB2024016
Record Dates: First submitted 2024-02-12; First posted 2024-02-29 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: High-Frequency Jet Ventilation; Bronchoscopy
MeSH Terms: interventions — High-Frequency Jet Ventilation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HFJV: All patients who underwent bronchoscopy with the use of high frequency jet ventilation between January 1st 2019 and december 31st 2023.
  Interventions: Procedure: High frequency jet ventilation

INTERVENTIONS:
Procedure: High frequency jet ventilation — Use of high frequency jet ventilation during bronchoscopy

SUMMARY:
High frequency jet ventilation (HFJV) has been introduced in 1967 as technique allowing ventilation with simultaneous access to the airway for bronchoscopy. Continuous improvement in the technique has led to a large use during interventional bronchoscopy, especially in large centers. However, complications occuring during the use of HFJV are poorly known. In this retrospective cohort study, the charts of all patients who had a bronchoscopy with the use of HFJV between 2019 and 2023 in our hospital will be analyzed. Primary outcome will the description of all complications during HFJV. Complications are defined as:

* Hypoxia: SpO2 < 90% for 1 min
* Severe hypoxia: SpO2 < 85% for 1 min
* Hemodynamic instability, defined as Arterial pressure < 90/60
* Cardiac arrhythmia
* Laryngospasm or bronchospasm
* Barotrauma or volutrauma
* Need for ICU admission

A model predicting the risk for developing any complication will be developped using 2 mathematical methods:

* a multivariate analysis
* a data mining approach

For both approaches, the following variables will be included in the model:

* Age
* Gender
* Weight
* Height
* BMI
* Smoking
* Alcohol consumption
* Consumption of Other drugs
* ASA class
* Obstructive pulmonary disease
* Restrictive lung disease
* COPD status (1, 2, 3, 4)
* Interstitial lung disease
* Lung tumor

  * Trachea location
  * Carina location
  * Bronchial location
* Pulmonary or tracheal stenosis
* Presence of stridor
* Severe stenosis (< 6 mm)
* Baseline SpO2 (pre-intervention)
* Pre-intervention oxygen requirement Procedure
* Duration (min)
* Stent placement
* Dilation
* Laser treatment
* Length of hospital stay Lung function tests
* FEV1 (forced expiratory volume)
* VC (Vital Capacity)
* FEV1/VC (Tiffeneau ratio)
* CPT (total lung capacity)
* DLCO (carbon monoxide diffusion)

ELIGIBILITY:
Inclusion Criteria:

* All patients who underwent a bronchoscopy with the use of high frequency jet ventilation between January 1st, 2019 and December 31st, 2023 at Erasme University Hospital, Brussels

Exclusion Criteria:

* Incomplete medical chart
* Patient who expressed their opposition to the use of their medical data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who underwent a bronchoscopy with the use of high frequency jet ventilation
Sampling Method: Non-Probability Sample
Enrollment: 1385 (Actual)
Dates: Start 2024-03-03 (Actual); Primary Completion 2024-03-19 (Actual); Study Completion 2025-02-01 (Actual)

PRIMARY OUTCOMES:
Occurence of complications | 6 hours
  The occurence (%) of complications of HFJV will be analyzed. Definition of complications is one or more of the following events:
  * Hypoxia: SpO2 < 90% for 1 min (%)
  * Severe hypoxia: SpO2 < 85% for 1 min (%)
  * Hemodynamic instability, defined as Arterial pressure < 90/60 (%)
  * Cardiac arrhythmia (%)
  * Laryngospasm or bronchospasm (%)
  * Barotrauma or volutrauma (%)
  * Need for ICU admission (%)
  Complications will be reported as overall complications (%) defined as the occurence of one or more of the listed events.
  Frequency of single events will be reported separately (%). Descriptive statistics ( %, mean, standard deviation, median, interquartile range) will be used as appropriate.

SECONDARY OUTCOMES:
Prediction model of complications | 6 hours
  A model predicting the risk for developing any complication will be developped using 2 mathematical methods:
  * a multivariate analysis
  * a data mining approach

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Universitaire de Bruxelles - Hôpital erasme, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aravena C, Mehta AC, Almeida FA, Lamb C, Maldonado F, Gildea TR. Innovation in rigid bronchoscopy-past, present, and future. J Thorac Dis. 2023 May 30;15(5):2836-2847. doi: 10.21037/jtd-22-779. Epub 2023 Apr 25. PMID 37324083
- [Background] Putz L, Mayne A, Dincq AS. Jet Ventilation during Rigid Bronchoscopy in Adults: A Focused Review. Biomed Res Int. 2016;2016:4234861. doi: 10.1155/2016/4234861. Epub 2016 Oct 26. PMID 27847813
- [Background] Poling HE, Wolfson B, Siker ES. A technique of ventilation during laryngoscopy and bronchoscopy. Br J Anaesth. 1975 Mar;47(3):382-4. doi: 10.1093/bja/47.3.382. PMID 1138745
- [Background] Klain M, Smith RB. High frequency percutaneous transtracheal jet ventilation. Crit Care Med. 1977 Nov-Dec;5(6):280-7. doi: 10.1097/00003246-197711000-00007. No abstract available. PMID 338247
- [Background] Hautmann H, Gamarra F, Henke M, Diehm S, Huber RM. High frequency jet ventilation in interventional fiberoptic bronchoscopy. Anesth Analg. 2000 Jun;90(6):1436-40. doi: 10.1097/00000539-200006000-00034. PMID 10825336
- [Background] Ost DE, Ernst A, Grosu HB, Lei X, Diaz-Mendoza J, Slade M, Gildea TR, Machuzak M, Jimenez CA, Toth J, Kovitz KL, Ray C, Greenhill S, Casal RF, Almeida FA, Wahidi M, Eapen GA, Yarmus LB, Morice RC, Benzaquen S, Tremblay A, Simoff M; AQuIRE Bronchoscopy Registry. Complications Following Therapeutic Bronchoscopy for Malignant Central Airway Obstruction: Results of the AQuIRE Registry. Chest. 2015 Aug;148(2):450-471. doi: 10.1378/chest.14-1530. PMID 25741903
- [Background] Goudra BG, Singh PM, Borle A, Farid N, Harris K. Anesthesia for Advanced Bronchoscopic Procedures: State-of-the-Art Review. Lung. 2015 Aug;193(4):453-65. doi: 10.1007/s00408-015-9733-7. Epub 2015 Apr 29. PMID 25921014
- [Background] Fernandez-Bustamante A, Ibanez V, Alfaro JJ, de Miguel E, German MJ, Mayo A, Jimeno A, Perez-Cerda F, Escribano PM. High-frequency jet ventilation in interventional bronchoscopy: factors with predictive value on high-frequency jet ventilation complications. J Clin Anesth. 2006 Aug;18(5):349-56. doi: 10.1016/j.jclinane.2005.12.011. PMID 16905080